CLINICAL TRIAL: NCT07105618
Title: Comparison of Dexmedetomidine Versus Fentanyl or Magnesium Sulphate as Adjuncts to Propofol-Based Total Intravenous Anesthesia in Patients Undergoing Craniotomy
Brief Title: Total Intravenous Anesthesia in Patients Undergoing Craniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Craniotomy anesthesia
Record Dates: First submitted 2025-07-08; First posted 2025-08-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Magnesium; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine group (Active Comparator): Intravenous loading dose of dexmedetomidine 1 µg/kg over 10 minutes before propofol infusion, followed by an intraoperative maintenance infusion of 0.5 µg/kg/hour.
  Interventions: Drug: Dexmedetomidine
- Fentanyl group (Active Comparator): Intravenous loading dose of fentanyl 1 µg/kg over 10 minutes before propofol infusion, followed by an intraoperative maintenance infusion of 0.5 µg/kg/hour.
  Interventions: Drug: Fentanyl
- Magnesium group (Active Comparator): Magnesium sulphate 30-50 mg/kg intravenous over 15-30 minutes before propofol infusion, followed by intraoperative maintenance infusion of 10-20 mg/kg/hour.
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine as an adjunct to total intravenous anesthesia.
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Fentanyl — Fentanyl as an adjunct to total intravenous anesthesia.
  Arms: Fentanyl group
Drug: Magnesium — Magnesium sulphate as an adjunct to total intravenous anesthesia.
  Other Names: Magnesium sulphate
  Arms: Magnesium group

SUMMARY:
Craniotomy presents true anesthetic challenges, mainly due to the need to optimize cerebral perfusion, facilitate brain relaxation, achieve rapid emergence for neurologic assessment, and minimize perioperative complications.

DETAILED DESCRIPTION:
Total intravenous anesthesia, particularly with propofol-based regimens, has gained favor in neurosurgical procedures for its neuroprotective properties, and reduced intracranial pressure; however, the choice of adjunct agents in total intravenous anesthesia remains a subject of ongoing investigation, especially regarding their influence on hemodynamic stability, analgesia, brain relaxation, and postoperative outcomes.

Total intravenous anesthesia techniques for craniotomy allow rapid recovery and stable hemodynamic parameters, so they decrease the hospital stay. The current study will compare the efficacy and safety profiles of dexmedetomidine, fentanyl, and magnesium sulfate as adjuncts in total intravenous anesthesia for patients undergoing craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Physical status: American Society of Anesthesiologists Physical Status (ASA) 1& II.
* Body mass index ≤ 30 kg/m2.
* Type of operation: elective craniotomy for brain tumor resection.
* Duration of surgery: within 4 hours.

Exclusion Criteria:

* Patient with hemodynamic instability or anticipated postoperative mechanical ventilation.
* Patients with a known history of allergy to the study drugs.
* Advanced hepatic, renal, cardiovascular, and neurologic diseases.
* Patients with chronic opioid use.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The total intraoperative propofol consumption | 4 hours
  The total intraoperative propofol consumption (in milligrams).

SECONDARY OUTCOMES:
Intraoperative heart rate | 4 hours
  Monitoring the changes in heart rate intraoperative.
Intraoperative mean arterial pressure | 4 hours
  Monitoring the changes in mean arterial pressure intraoperative.
Additional doses of intraoperative fentanyl. | 4 hours
  The total number of patients requiring additional dose of intraoperative fentanyl.
The time to first request for rescue analgesia | The first 24 hours postoperative.
  The time to first request for rescue analgesia in first 24 hour.
Postoperative pain assessment | The first 24 hours postoperative.
  Postoperative pain assessment by the numeric rating scale in the recovery room and at 2,4,8,16 and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mahmoud Ahmed, MD, Principal Investigator — Department of Anesthesia, Intensive Care & Pain Management, Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Egypt

REFERENCES:
- [Background] Ali AR, El Ghoneimy MN. Dexmedetomidine versus fentanyl as adjuvant to propofol: comparative study in children undergoing extracorporeal shock wave lithotripsy. Eur J Anaesthesiol. 2010 Dec;27(12):1058-64. doi: 10.1097/EJA.0b013e32833e6e2d. PMID 20805754
- [Background] Telci L, Esen F, Akcora D, Erden T, Canbolat AT, Akpir K. Evaluation of effects of magnesium sulphate in reducing intraoperative anaesthetic requirements. Br J Anaesth. 2002 Oct;89(4):594-8. doi: 10.1093/bja/aef238. PMID 12393361
- [Background] Chandar Chinnarasan V, Bidkar PU, Swaminathan S, Mani M, Vairappan B, Chatterjee P, Joy JJ, Dey A, Ramadurai R, Gunasekaran A. Comparison of dexmedetomidine versus fentanyl-based total intravenous anesthesia technique on the requirement of propofol, brain relaxation, intracranial pressure, neuronal injury, and hemodynamic parameters in patients with acute traumatic subdural hematoma undergoing emergency craniotomy: A randomized controlled trial. Surg Neurol Int. 2024 Dec 13;15:462. doi: 10.25259/SNI_892_2024. eCollection 2024. PMID 39777171
- [Background] Preethi J, Bidkar PU, Cherian A, Dey A, Srinivasan S, Adinarayanan S, Ramesh AS. Comparison of total intravenous anesthesia vs. inhalational anesthesia on brain relaxation, intracranial pressure, and hemodynamics in patients with acute subdural hematoma undergoing emergency craniotomy: a randomized control trial. Eur J Trauma Emerg Surg. 2021 Jun;47(3):831-837. doi: 10.1007/s00068-019-01249-4. Epub 2019 Oct 29. PMID 31664468